CLINICAL TRIAL: NCT01292317
Title: Early Detection and Intervention of Acute Contrast Media Induced Nephropathy Using Neutrophil Gelatinase-associated Lipocalin (NGAL) May Improve Renal Outcome: A Study in Patients Undergoing Intra-arterial Angiography.
Brief Title: Neutrophil Gelatinase-associated Lipocalin (NGAL) and Contrast Media Induced Nephropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Abbott Diagnostics Division (Industry)
Responsible Party: Principal Investigator, Gernot Schilcher, MD, Joerg Horina, Professor of Medicine, Medical University of Graz, Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CIN and NGAL 1.0; Ek 21-278 ex 09/10 (Other: Ethics Committee Medical University Graz)
Record Dates: First submitted 2011-02-08; First posted 2011-02-09 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Contrast Media Induced Nephropathy (CIN)
Keywords: NGAL; neutrophil gelatinase-associated Lipocalin; contrast media nephropathy; CIN; volume expansion; acute kidney injury; contrast media
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous hydration (Active Comparator): intravenous application of 0.9% saline
  Interventions: Other: application of intravenous volume
- oral hydration only (Active Comparator)
  Interventions: Other: oral fluid application

INTERVENTIONS:
Other: application of intravenous volume — weight based intravenous application of volume
  Arms: intravenous hydration
Other: oral fluid application — oral fluid application
  Arms: oral hydration only

SUMMARY:
Introduction:

Patients with pre-existing impaired renal function are prone to develop acute contrast media induced nephropathy (CIN). Neutrophil gelatinase-associated Lipocalin (NGAL), a new biomarker predictive for acute renal injury has been shown to be capable for earlier diagnosis of acute contrast media induced nephropathy (CIN) in patients undergoing cardiac surgery.

Intravenous volume load is a widely accepted prophylaxis.

In this randomized and controlled study, only patients with the need for an intra-arterial contrast media (CM) application will be included and receive a standardized, weight-based, intravenous hydration before investigation.

It is the aim of this study:

1. to evaluate the magnitude of a risk for contrast media induced nephropathy (CIN) following intra-arterial angiography in a well defined group of high-risk patients.
2. to use urinary Neutrophil gelatinase-associated Lipocalin (NGAL) as an early predictor of contrast media induced nephropathy (CIN) after contrast media (CM) application.
3. to evaluate the clinical benefit of an early post-procedural i.v. hydration as compared to only pre-procedural volume expansion.

Patients with markedly increased urinary Neutrophil gelatinase-associated Lipocalin (NGAL) after investigation will be randomized into one of two study groups:

Patients of Group A will undergo standard treatment consisting of unrestricted oral fluid intake.

Patients of Group B will additionally receive 3-4 ml/kg BW/h 0.9 % saline intravenously for 6 hours.

Endpoints:

Primary endpoint: contrast media induced nephropathy (CIN) defined by an increase greater than 25% of baseline serum creatinine.

Secondary endpoint: NGAL, Cystatin C, and creatinine values, need for renal replacement therapy, death.

DETAILED DESCRIPTION:
Introduction:

Over the last decades the growing demand for appropriate diagnosing and intervention in all fields of modern medicine has increased the necessity for use of iodinated contrast media (CM). Patients with pre-existing impaired renal function are prone to develop acute contrast media induced nephropathy (CIN) and consecutively have a greater risk of death.

To date, a reliable laboratory value or test that recognizes acute renal damage before serum creatinine increases is still sought for. It would be a most helpful tool to initiate proper treatment on time. Neutrophil gelatinase-associated Lipocalin (NGAL), a new biomarker predictive for acute renal injury has been shown to be capable for earlier diagnosis of contrast media induced nephropathy (CIN) in patients undergoing cardiac surgery.

So far, an intravenous volume load is the only fairly proven and widely accepted prophylaxis. However, the optimal intravenous fluid regimen regarding the type, amount, route and duration of volume application has remained controversial. Habits of giving pre- and post-procedural volume have been widely differing throughout all randomized trials and, thus, are not comparable in the available studies. Unfortunately, most studies were also lacking statistical power, used different types of contrast media (CM) and definitions of contrast media induced nephropathy (CIN) or allowed for additional prophylactic measures, such as N-acetylcysteine or sodium bicarbonate in a varying percentage of their patients.

In our randomized and controlled study, only patients with the need for an intra-arterial contrast media (CM) application will be included. Patients scheduled for a diagnostic angiography and/or endovascular intervention will receive a standardized, weight-based, intravenous hydration before investigation. Only one type of contrast media (CM) and neither sodium bicarbonate, nor N-acetylcysteine is used throughout the study. The study will be performed according to the Consort-Statement 2010 for clinical trials.

It is the aim of our study:

1. to evaluate the magnitude of a risk for contrast media induced nephropathy (CIN) following intra-arterial angiography in a well defined group of high-risk patients.
2. to use urinary Neutrophil gelatinase-associated Lipocalin (NGAL) as an early predictor of contrast media induced nephropathy (CIN) after contrast media (CM) application.
3. to evaluate the clinical benefit of an early post-procedural i.v. hydration as compared to only pre-procedural volume expansion.

Patients with markedly increased Neutrophil gelatinase-associated Lipocalin (NGAL) values (criteria for randomization into one of two treatment groups see below) at 4 to 6 hours after investigation will be randomized into one of two study groups:

Patients of Group A will additionally receive 3-4 ml/kg BW/h 0.9 % saline intravenously for 6 hours.

Patients of Group B will undergo standard treatment consisting of unrestricted oral fluid intake, at least 500 ml tea or water provided by the ward, but no intravenous fluid application.

Criteria for Randomization (after 2nd NGAL testing):

* Patients with NGAL levels > 150 ng/ml, if baseline was below 75 ng/ml.
* Patients with doubling of NGAL values, if baseline was between 75 and 150 ng/ml.

Endpoints:

Primary endpoint: contrast media induced nephropathy (CIN) defined by an increase greater than 25% of baseline serum creatinine.

Secondary endpoint: NGAL, Cystatin C, and creatinine values, need for renal replacement therapy, death.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the need for intra-arterial angiography/angioplasty
* Patients older than 18 years
* Patients with clinically stable chronic renal insufficiency stage 2 and more (calculated GFR < 70 ml/min/1,73 m2)(65)
* Written informed consent

Exclusion Criteria:

* Pre-existing clinical and/or laboratory evidence of acute renal failure at the time of enrollment
* Evidence of rhabdomyolysis
* Patients on renal replacement therapy (34)
* Patients with life-threatening underlying disease (sepsis, MOF, SIRS)
* Contraindication for volume therapy
* Pregnancy
* Contrast media application within 7 days prior to intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 819 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Contrast media induced nephropathy (CIN) defined by an increase greater than 25% of baseline serum creatinine. | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Horina, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Medicine, Division of Nephrology, Graz, Styria, Austria

REFERENCES:
- [Background] Reddan D, Laville M, Garovic VD. Contrast-induced nephropathy and its prevention: What do we really know from evidence-based findings? J Nephrol. 2009 May-Jun;22(3):333-51. PMID 19557710
- [Background] Haase-Fielitz A, Bellomo R, Devarajan P, Story D, Matalanis G, Dragun D, Haase M. Novel and conventional serum biomarkers predicting acute kidney injury in adult cardiac surgery--a prospective cohort study. Crit Care Med. 2009 Feb;37(2):553-60. doi: 10.1097/CCM.0b013e318195846e. PMID 19114878
- [Background] McCullough PA, Wolyn R, Rocher LL, Levin RN, O'Neill WW. Acute renal failure after coronary intervention: incidence, risk factors, and relationship to mortality. Am J Med. 1997 Nov;103(5):368-75. doi: 10.1016/s0002-9343(97)00150-2. PMID 9375704
- [Derived] Ribitsch W, Schilcher G, Quehenberger F, Pilz S, Portugaller RH, Truschnig-Wilders M, Zweiker R, Brodmann M, Stiegler P, Rosenkranz AR, Pickering JW, Horina JH. Neutrophil gelatinase-associated lipocalin (NGAL) fails as an early predictor of contrast induced nephropathy in chronic kidney disease (ANTI-CI-AKI study). Sci Rep. 2017 Jan 27;7:41300. doi: 10.1038/srep41300. PMID 28128223
- [Derived] Schilcher G, Ribitsch W, Otto R, Portugaller RH, Quehenberger F, Truschnig-Wilders M, Zweiker R, Stiegler P, Brodmann M, Weinhandl K, Horina JH. Early detection and intervention using neutrophil gelatinase-associated lipocalin (NGAL) may improve renal outcome of acute contrast media induced nephropathy: a randomized controlled trial in patients undergoing intra-arterial angiography (ANTI-CIN Study). BMC Nephrol. 2011 Aug 17;12:39. doi: 10.1186/1471-2369-12-39. PMID 21849080